CLINICAL TRIAL: NCT00443391
Title: The Long-Term Safety and Tolerability of ABT-089 in Adults With Attention Deficit-Hyperactivity Disorder (ADHD): An Open-Label Extension Study
Brief Title: A Safety and Tolerability Study of ABT-089 in Adults With Attention Deficit-Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-889
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — pozanicline

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABT-089

INTERVENTIONS:
Drug: ABT-089 — Open label study, subjects will take up to 80mg daily for 24 months.

SUMMARY:
The objective of this study is to evaluate the long-term safety and tolerability of ABT-089 in adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* The subject was randomized into Study M06-855 and completed treatment in Periods 1 and 2 and the 2-week Extension Period
* If female, subject must be either postmenopausal for at least 1 year, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or practicing at least a method of birth control throughout the study
* If female, the result of a pregnancy tests are negative
* The subject is judged to be in generally good health

Exclusion Criteria:

* More than 7 days have elapsed since the last dose of study drug in Study M06-855
* The subject has taken any ADHD medication between the last dose of study drug in Study M06-855 and the first dose of study drug in the current study
* The subject anticipates a move outside the geographic area

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
CAARS:INV | Day -1, Day 14, Months 1, 2, 3, 6, 9, 12, 15, 18, 21, 24
CGI-ADHD-S | Day -1, Day 14, Months 1, 2, 3, 6, 9, 12, 15, 18, 21, 24

SECONDARY OUTCOMES:
AAQoL | Day -1, Months 3, 6, 9, 12, 15, 18, 21, 24
WPAI | Day -1, Months 3, 6, 9, 12, 15, 18, 21, 24
RUQ | Day -1, Months 3, 6, 9, 12, 15, 18, 21, 24
FTND | Day -1, Months 1, 2, 3, 6, 9, 12, 15, 18, 21, 24

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, MD, PhD, MD, Study Director — AbbVie
Locations (21):
- United States (21):
  - Site Reference ID/Investigator# 6109, Mesa, Arizona
  - Site Reference ID/Investigator# 6765, Mesa, Arizona
  - Site Reference ID/Investigator# 6100, Lafayette, California
  - Site Reference ID/Investigator# 6107, San Diego, California
  - Site Reference ID/Investigator# 6112, Jacksonville, Florida
  - Site Reference ID/Investigator# 6096, Maitland, Florida
  - Site Reference ID/Investigator# 6105, Tampa, Florida
  - Site Reference ID/Investigator# 6094, Smyrna, Georgia
  - Site Reference ID/Investigator# 6111, Newton, Kansas
  - Site Reference ID/Investigator# 6113, Farmington Hills, Michigan
  - Site Reference ID/Investigator# 6110, Omaha, Nebraska
  - Site Reference ID/Investigator# 6099, New York, New York
  - Site Reference ID/Investigator# 6106, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 6102, Portland, Oregon
  - Site Reference ID/Investigator# 6097, Charleston, South Carolina
  - Site Reference ID/Investigator# 6098, Memphis, Tennessee
  - Site Reference ID/Investigator# 6103, Austin, Texas
  - Site Reference ID/Investigator# 6104, Lake Jackson, Texas
  - Site Reference ID/Investigator# 6095, Herndon, Virginia
  - Site Reference ID/Investigator# 6092, Seattle, Washington
  - Site Reference ID/Investigator# 6101, Middleton, Wisconsin